CLINICAL TRIAL: NCT03971903
Title: Department of Psychology, Hunan Normal University
Brief Title: Attention Bias Modification Treatment for Young Adults With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Wenhui Yang, Department of Psychology, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBA130016
Record Dates: First submitted 2018-01-31; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Depressive Disorder, Major
Keywords: Attenion bias modification, major depression, treatment
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Particpants are assigned to active ABM treatment or placebo training
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention bias modification treatment (Experimental): 12-session of ABMT
  Interventions: Behavioral: Attention bias modification
- Placebo controls (Placebo Comparator): 12-session of placebo(i.e.,sham) training
  Interventions: Behavioral: Attention bias modification

INTERVENTIONS:
Behavioral: Attention bias modification — The ABM training task was a variation of the computerized visual dot-probe task. During the training, each session includes 54 neutral-sad word pairs presenting 6 times (6 × 54=324 trials) during 20-minute. Participants received 12 sessions over 4 weeks (1 session every other day). In the active ABMT, 90% of the probes appeared at the neutral position and 10% at the sad position. At the placebo ABMT, 50% of the probes appeared at the neutral position and 50% at the sad position.

SUMMARY:
In this study, the investigators test whether a 4-week 12-session attention bias modification treatment (ABMT) could reduce depressive symptoms relative to placebo controls in young adults with major depressive disorder at post-training and 3-month follow-ups. Meanwhile, the investigators also test whether a 2-week 4-session ABMT booster training for every three months could reduce residual depressive symptoms and recurrences relative to placebo controls for 1-year follow-up

DETAILED DESCRIPTION:
Attention Bias Modification Training was a modified dot-probe task, in which 90% of the targets appeared at the neutral word position and 10% at the sad word position. The placebo training procedure is a classic dot-probe task in which the targets appeared with equal probability in the sad (50%) and neutral (50%) word positions. The investigators assess attention bias scores, depressive symptoms, trait anxiety, rumination and self-report attention control ability at 1-week, 2-week, 4-week,7-week,3-month,4-month, 5-month, 6-month and 12-month follow-ups after training.

ELIGIBILITY:
Inclusion Criteria:

* The presence of definite and probable MDD (i.e., at least 1 core symptom plus 3 further depressive symptoms present for at least 2 weeks) diagnoses

Exclusion Criteria:

* a diagnosis of bipolar disorder, schizophrenia, or mood disorder due to a general medical condition or substance-induced mood disorder; and any concurrent treatment (i.e., psychotherapy and/or pharmacotherapy).

Ages: 16 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2017-12-24 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Changes of attention bias score | pre-training, post-training(4 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month(booster pre-training),4-month(booster post-training),5-month,6-month,12-month after post-training )
  Attention bias score changes tested by a typical dot-probe task
Changes of depressive symptoms | pre-training, post-training(4 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month(booster pre-training),4-month(booster post-training),5-month,6-month,12-month after post-training )
  Depression symptoms tested by clinicians using Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS)
Changes of severity of depression | pre-training, post-training(4 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month(booster pre-training),4-month(booster post-training),5-month,6-month,12-month after post-training )
  The severity of depression tested by clinicians using the 17-Item Hamilton Depression Rating Scale (HAM-D)

SECONDARY OUTCOMES:
Changes of self-reported depressive symptoms | pre-training, post-training(4 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month(booster pre-training),4-month(booster post-training),5-month,6-month,12-month after post-training )
  Self-reported depressive symptoms assessed by Beck depression scale-second version (BDI-II), and trait anxiety assessed by State Trait Anxiety Inventory-Trait(STAI-T), rumination assessed by Rumination Response Scale(RRS).
Changes of self-reported trait anxiety | pre-training, post-training(4 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month(booster pre-training),4-month(booster post-training),5-month,6-month,12-month after post-training )
  self-reported trait anxiety assessed by State Trait Anxiety Inventory-Trait(STAI-T)
Changes of self-reported rumination | pre-training, post-training(4 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month(booster pre-training),4-month(booster post-training),5-month,6-month,12-month after post-training )
  Self-reported rumination assessed by Rumination Response Scale(RRS).

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Yang, Ph.D, Principal Investigator — Hunan Normal University
Locations (1):
- Department of Psychology, Hunan Normal University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
After completion, all the data can be shared
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After 2020 and forever
Access Criteria: Just for research

REFERENCES:
- [Background] Yang W, Ding Z, Dai T, Peng F, Zhang JX. Attention Bias Modification training in individuals with depressive symptoms: A randomized controlled trial. J Behav Ther Exp Psychiatry. 2015 Dec;49(Pt A):101-11. doi: 10.1016/j.jbtep.2014.08.005. Epub 2014 Sep 8. PMID 25245928
- [Result] Yang W, Zhang JX, Ding Z, Xiao L. Attention Bias Modification Treatment for Adolescents With Major Depression: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2016 Mar;55(3):208-18.e2. doi: 10.1016/j.jaac.2015.12.005. Epub 2015 Dec 23. PMID 26903254